CLINICAL TRIAL: NCT04115189
Title: A Retrospective Medical Record Review of First-Line Sunitinib Administration Schedules and Outcomes Among Patients With Metastatic Renal Cell Carcinoma in Latin America
Brief Title: A Retrospective Medical Record Review of First-Line Sunitinib Administration Schedules and Outcomes Among Patients With mRCC in Latin America (LA)
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A6181231
Record Dates: First submitted 2019-10-02; First posted 2019-10-03 (Actual); Results first posted 2022-05-10 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2022-02

CONDITIONS: Metastatic Renal Cell Carcinoma ( mRCC)
Keywords: Sunitinib -
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Sunitinib

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with Metastatic RCC: Patients diagnosed with metastatic RCC with clear cell histology who switched from a 4/2 schedule to a 2/1 schedule of sunitinib in first-line metastatic treatment between January 1, 2014 and June 30, 2018
  Interventions: Drug: Sunitinib

INTERVENTIONS:
Drug: Sunitinib — Patients to receive Sunitinib as first line therapy for mRCC

SUMMARY:
To describe real-world demographic and clinical characteristics, treatment characteristics, and clinical outcomes among patients in Latin America who were treated with first-line sunitinib for metastatic renal cell carcinoma and switched from the 4/2 to 2/1 administration schedule

DETAILED DESCRIPTION:
Understanding characteristics of patients who switched from a 4/2 to a 2/1 sunitinib schedule or initiated the 2/1 schedule in Brazil, and the resulting clinical outcomes in the real-world setting

• Describing the occurrence of AEs on the 4/2 and 2/1 schedules

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with metastatic RCC with clear cell histology

   a. The patient may have been initially diagnosed with Stage IV or initially diagnosed at an earlier stage and progressed to having disease at distant sites (i.e., metastatic disease)
2. Initiated first-line treatment for metastatic RCC with sunitinib on the 4/2 schedule (all countries) or initiated first-line treatment for metastatic RCC with sunitinib on the 2/1 schedule (Brazil only)
3. Switched to the 2/1 schedule (all countries) or initiated the 2/1 schedule (Brazil only) during the first treatment line between January 1, 2014, and June 30, 2018 a. The final dates defining this selection period will be dependent on country-specific ethics and reporting requirements

Exclusion Criteria:

1. Evidence of other malignant neoplasms (except nonmelanoma skin cancer or carcinoma in situ) within 5 years before switching to the sunitinib 2/1 schedule (all countries) or initiation of the 2/1 schedule (Brazil only)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with clear cell mRCC at age 18 or older who initiated sunitinib as first-line treatment between 2014-2018
Sampling Method: Non-Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2019-12-13 (Actual); Primary Completion 2020-12-02 (Actual); Study Completion 2020-12-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (7):
- Argentina (3):
  - Instituto Médico Especializado Alexander Fleming, Buenos Aires
  - Sanatorio del Salvador - Cordoba, Córdoba
  - Centro Oncológico de Integración Regional in Mendoza, Mendoza
- Escola Paulista de Medicina - UNIFESP, São Paulo, Brazil
- Colombia (2):
  - Fundacion Cardiovascular de Colombia, Bogotá
  - Sociedad de Oncologia y Hematologia Del Cesar ltda (SOHEC), Valledupar
- Hospital Eugenio Espejo, Quito, Ecuador

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=A6181231

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who were diagnosed with metastatic renal cell carcinoma (mRCC), as per customized retrospective medical record review conducted in 7 countries (Argentina, Brazil, Colombia, Costa Rica, Ecuador, Mexico, and Peru) from January 2014 to June 2018 (+/- 6 months, maximum up to 5 years), and treated with Sunitinib, were included in this study and their data was observed retrospectively.
Pre-assignment Details: The index date was the date of switching first-line treatment from 4/2 administration schedule (4 weeks sunitinib treatment followed by 2 weeks off treatment) to 2/1 administration schedule (2 weeks sunitinib treatment followed by 1 week off treatment) or initiating first-line treatment on the 2/1 schedule.
Groups:
- Sunitinib: Switched From 4/2 to 2/1 Schedule: Participants with mRCC who initiated first-line treatment with sunitinib 50 mg per day on 4/2 schedule then switched to 2/1 schedule in the daily clinical practice, between 1-Jan-2014 and 30-Jun-2018 (+/- 6 months) were observed retrospectively over a duration of approximately 12 months.
- Sunitinib 2/1 Schedule: Participants with mRCC who initiated first-line treatment with sunitinib 50 mg on 2/1 schedule in the daily clinical practice, between 1-Jan-2014 and 30-Jun-2018 (+/- 6 months), were observed retrospectively over a duration of approximately 12 months.
Period: Overall Study
Arm/Group | Sunitinib: Switched From 4/2 to 2/1 Schedule | Sunitinib 2/1 Schedule
Started | 42 | 15
Completed | 42 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Analysis population included all eligible participants whose data were retrieved from medical records and studied.
Groups:
- Total: Total of all reporting groups
Arm/Group | Sunitinib: Switched From 4/2 to 2/1 Schedule | Sunitinib 2/1 Schedule | Total
Number analyzed (Participants) | 42 | 15 | 57
Age, Customized [Count of Participants; unit: Participants]
  18 to 39 years | 1 | 1 | 2
  40 to 49 years | 6 | 1 | 7
  50 to 59 years | 15 | 6 | 21
  60 to 69 years | 15 | 4 | 19
  >=70 years | 5 | 0 | 5
  Unknown | 0 | 3 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 3 | 26
  Male | 19 | 12 | 31
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Demographic Characteristic of Participants: Year of Birth
Time Frame: During pre-index period (anytime from initial metastatic diagnosis to before index date), during data identification period of 5 years (data recorded during approximately 12 months of retrospective observation period)
Population: Analysis population included all eligible participants whose data were retrieved from medical records and assessed.
Measure: Count of Participants; unit: Participants
Arm/Group | Sunitinib: Switched From 4/2 to 2/1 Schedule | Sunitinib 2/1 Schedule
Number analyzed (Participants) | 42 | 15
Participants
  Year: 1937 | 1 | 0
  Year: 1939 | 1 | 0
  Year: 1942 | 1 | 0
  Year: 1943 | 1 | 0
  Year: 1944 | 1 | 2
  Year: 1946 | 1 | 1
  Year: 1947 | 2 | 1
  Year: 1948 | 2 | 0
  Year: 1949 | 1 | 0
  Year: 1950 | 2 | 0
  Year: 1951 | 2 | 1
  Year: 1952 | 2 | 0
  Year: 1953 | 5 | 0
  Year: 1954 | 2 | 0
  Year: 1955 | 2 | 0
  Year: 1956 | 1 | 2
  Year: 1957 | 4 | 1
  Year: 1958 | 2 | 2
  Year: 1959 | 2 | 0
  Year: 1960 | 0 | 1
  Year: 1963 | 1 | 2
  Year: 1965 | 1 | 0
  Year: 1966 | 1 | 0
  Year: 1968 | 0 | 1
  Year: 1969 | 2 | 0
  Year: 1975 | 1 | 0
  Year: 1978 | 1 | 0
  Year: 1983 | 0 | 1

2. Primary Outcome: Demographic Characteristic of Participants: Comorbidities
Description: Data for participants with following comorbidities were observed and reported: cerebrovascular disease,chronic pulmonary disease,congestive heart failure,connective tissue disease,dementia,diabetes with end organ damage,diabetes without end organ damage,depression,hemiplegia or paraplegia, history of myocardial infarction,human immunodeficiency virus/ acquired immunodeficiency syndrome,hypertension,mild liver disease (i.e., chronic hepatitis or cirrhosis without portal hypertension),moderate to severe liver disease (i.e., cirrhosis and portal hypertension),use of warfarin,moderate to severe renal disease (i.e., creatinine >3mg% [265 mcmol/l],dialysis,transplantation,uremic syndrome),ulcer disease,peripheral vascular disease,skin ulcers/cellulitis,horseshoe kidney,polycystic kidney disease,von hippel-lindau disease,chronic viral hepatitis, previous thyroid disorders. Categories with at least 1 non-zero data are reported below. One participant could have more than 1 comorbidities.
Time Frame: as for outcome 1
Population: Analysis population included all eligible participants whose data were retrieved from medical records and assessed.
Measure: Count of Participants; unit: Participants
Arm/Group | Sunitinib: Switched From 4/2 to 2/1 Schedule | Sunitinib 2/1 Schedule
Number analyzed (Participants) | 42 | 15
Participants
  Cerebrovascular disease | 1 | 0
  Congestive heart failure | 1 | 1
  Diabetes with end organ damage | 3 | 0
  Diabetes without end organ damage | 7 | 5
  Depression | 3 | 0
  History of myocardial infarction | 4 | 0
  Hypertension | 27 | 10
  Mild liver disease | 1 | 0
  Moderate to severe renal disease | 2 | 0
  Horseshoe kidney | 0 | 1
  Polycystic kidney disease | 0 | 1
  Previous thyroid disorders | 5 | 0

3. Primary Outcome: Demographic Characteristic of Participants: Primary Health Insurance Type
Description: Participants with following insurance status were observed and reported: Private insurance only and public insurance.
Time Frame: as for outcome 1
Population: Analysis population included all eligible participants whose data were retrieved from medical records and assessed.
Measure: Count of Participants; unit: Participants
Arm/Group | Sunitinib: Switched From 4/2 to 2/1 Schedule | Sunitinib 2/1 Schedule
Number analyzed (Participants) | 42 | 15
Participants
  Public health plan | 11 | 7
  Private health plan | 31 | 6
  Unknown | 0 | 2

4. Primary Outcome: Demographic Characteristic of Participants: Height
Time Frame: as for outcome 1
Population: Analysis population included all eligible participants whose data were retrieved from medical records and assessed. Here, 'overall number of participants analyzed' signifies number of participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Centimeter
Arm/Group | Sunitinib: Switched From 4/2 to 2/1 Schedule | Sunitinib 2/1 Schedule
Number analyzed (Participants) | 21 | 8
Centimeter | 164.4 (10.4) | 168.9 (6.6)

5. Primary Outcome: Demographic Characteristic of Participants: Weight
Time Frame: as for outcome 1
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Kilograms
Arm/Group | Sunitinib: Switched From 4/2 to 2/1 Schedule | Sunitinib 2/1 Schedule
Number analyzed (Participants) | 28 | 8
Kilograms | 73.5 (13.6) | 90.5 (12.4)

6. Primary Outcome: Demographic Characteristic of Participants: Body Mass Index
Description: Body mass index (BMI) is calculated as the body mass in kilograms divided by the square of the body height in meters.
Time Frame: as for outcome 1
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Kilogram per square meter (kg/m^2)
Arm/Group | Sunitinib: Switched From 4/2 to 2/1 Schedule | Sunitinib 2/1 Schedule
Number analyzed (Participants) | 21 | 8
Kilogram per square meter (kg/m^2) | 28.2 (5.7) | 31.8 (4.4)

7. Primary Outcome: Clinical Characteristic of Participants: Year of Diagnosis of Metastatic Renal Cell Carcinoma
Description: In this outcome measure participants diagnosed with mRCC between 2012 to 2018 were reported.
Time Frame: as for outcome 1
Population: Analysis population included all eligible participants whose data were retrieved from medical records and assessed.
Measure: Count of Participants; unit: Participants
Arm/Group | Sunitinib: Switched From 4/2 to 2/1 Schedule | Sunitinib 2/1 Schedule
Number analyzed (Participants) | 42 | 15
Participants
  Year: 2012 | 1 | 0
  Year: 2013 | 2 | 1
  Year: 2014 | 3 | 0
  Year: 2015 | 9 | 1
  Year: 2016 | 8 | 5
  Year: 2017 | 15 | 4
  Year: 2018 | 4 | 3
  Unknown | 0 | 1

8. Primary Outcome: Clinical Characteristic of Participants: Stages of Renal Cell Carcinoma (RCC)
Description: The American Joint Committee on Cancer (AJCC) stages were assigned. Stage I- defined as tumor of 7 cm across or smaller, while Stage II- defined as tumor larger than 7 cm across and did not spread to lymph nodes or distant organs, Stage III- defined as tumor was growing into a major vein (like the renal vein or the vena cava) or into tissue around the kidney, but it was not growing into the adrenal gland or beyond Gerota's fascia. There was no spread to lymph nodes or distant organs. Stage IV- defined as main tumor was growing beyond Gerota's fascia and may be growing into the adrenal gland on top of the kidney. It might or might not had spread to nearby lymph nodes. It had not spread to distant lymph nodes or other organs.
Time Frame: as for outcome 1
Population: Analysis population included all eligible participants whose data were retrieved from medical records and assessed.
Measure: Count of Participants; unit: Participants
Arm/Group | Sunitinib: Switched From 4/2 to 2/1 Schedule | Sunitinib 2/1 Schedule
Number analyzed (Participants) | 42 | 15
Participants
  Stage I | 1 | 0
  Stage II | 6 | 1
  Stage III | 6 | 1
  Stage IV | 17 | 10
  Unknown | 12 | 3

9. Primary Outcome: Clinical Characteristic of Participants: Risk Groups
Description: Participants with Memorial Sloan Kettering Cancer Center(MSKCC)model and International Metastatic Renal Cell Carcinoma Database Consortium(IMDC)criteria risks groups are reported.MSKCC model assessed as low(0),intermediate(1-2) or high risk(=>3)based on number of criteria present.Criteria=Karnofsky performance status(KPS)score <80,lactate dehydrogenase>1.5*upper limit of normal,hemoglobin<lower limit of normal, corrected serum calcium>10 mg/dL,time from first diagnosis of RCC to start of systemic therapy of<1 year.KPS score range:0=death to 100=no evidence of disease,higher score=higher ability to perform daily tasks.IMDC risk group stratifies participants in poor,intermediate(had 1 or 2 poor factors)and favorable(had no poor factors)risk groups based on number of adverse clinical,laboratory parameters.Poor factors included KPS score of<80 at initiation of treatment,time from diagnosis to metastasis treatment of<12 months,anemia,corrected calcium>10 mg/dL,neutrophilia,thrombocythemia.
Time Frame: as for outcome 1
Population: Analysis population included all eligible participants whose data were retrieved from medical records and assessed. Here, "number analyzed" signifies the number of participants evaluable at specific category.
Measure: Count of Participants; unit: Participants
Arm/Group | Sunitinib: Switched From 4/2 to 2/1 Schedule | Sunitinib 2/1 Schedule
Number analyzed (Participants) | 42 | 15
Participants
  MSKCC: Low risk | 25 | 6
  MSKCC: Intermediate risk | 12 | 7
  MSKCC: Poor risk | 5 | 2
  IMDC: Favorable risk: number analyzed (Participants) | 17 | 0
  IMDC: Favorable risk | 4 | 0
  IMDC: Intermediate risk: number analyzed (Participants) | 17 | 0
  IMDC: Intermediate risk | 11 | 0
  IMDC: Poor risk: number analyzed (Participants) | 17 | 0
  IMDC: Poor risk | 2 | 0

10. Primary Outcome: Clinical Characteristic of Participants: Sites of Distant Metastases
Description: Number of participants with the sites of distant metastasis at initial metastatic diagnosis are reported in this outcome measure. Sites evaluated for distant metastasis were lymph nodes, bone, brain, liver, lung/pleura, adrenal gland, pancreas, others (peritoneum, surgical lodge, soft tissue, nephrectomy bed). One participant could have more than 1 sites of metastases.
Time Frame: as for outcome 1
Population: Analysis population included all eligible participants whose data were retrieved from medical records and assessed.
Measure: Count of Participants; unit: Participants
Arm/Group | Sunitinib: Switched From 4/2 to 2/1 Schedule | Sunitinib 2/1 Schedule
Number analyzed (Participants) | 42 | 15
Participants
  Lymph nodes | 13 | 3
  Bone | 10 | 2
  Brain | 3 | 1
  Liver | 8 | 1
  Lung/pleura | 25 | 8
  Adrenal gland | 5 | 2
  Pancreas | 2 | 2
  Other: Peritoneum | 3 | 0
  Other: Surgical lodge | 2 | 0
  Other: Soft tissue | 2 | 0
  Other: Nephrectomy bed | 1 | 0

11. Primary Outcome: Clinical Characteristic of Participants: Eastern Cooperative Oncology Group (ECOG) Performance Status
Description: The ECOG performance status was used to assess the effect of disease progression on participant's daily activities. ECOG performance status Grade 0: fully active, able to carry on all pre-disease performance without restriction; Grade 1: restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, Grade 2: ambulatory and capable of all self-care, but unable to carry out any work activities, up and about more than 50% of waking hours, Grade 3: capable of only limited self-care, confined to bed or chair for more than 50% of waking hours, Grade 4: completely disabled; cannot carry on any self-care; totally confined to bed or chair.
Time Frame: as for outcome 1
Population: Analysis population included all eligible participants whose data were retrieved from medical records and assessed.
Measure: Count of Participants; unit: Participants
Arm/Group | Sunitinib: Switched From 4/2 to 2/1 Schedule | Sunitinib 2/1 Schedule
Number analyzed (Participants) | 42 | 15
Participants
  Grade 0 | 13 | 5
  Grade 1 | 23 | 7
  Grade 2 | 3 | 1
  Grade 3 | 0 | 0
  Grade 4 | 0 | 0
  Unknown | 3 | 2

12. Primary Outcome: Treatment Modalities Received Prior to Metastatic Renal Cell Carcinoma (mRCC) Diagnosis
Description: In this outcome measure participants with different treatment modalities including partial nephrectomy, radical nephrectomy, radiation therapy, neoadjuvant systemic therapy and adjuvant systemic therapy were reported. One participant could have more than 1 treatment modalities.
Time Frame: Before diagnosis of mRCC, anytime during data identification period of 5 years (data recorded during approximately 12 months of retrospective observation period)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Sunitinib: Switched From 4/2 to 2/1 Schedule | Sunitinib 2/1 Schedule
Number analyzed (Participants) | 28 | 9
Participants
  Partial nephrectomy | 1 | 0
  Radical nephrectomy | 28 | 8
  Radiation therapy | 0 | 0
  Neoadjuvant systemic therapy | 0 | 1
  Adjuvant systemic therapy | 0 | 0

13. Primary Outcome: Duration Between Last Treatment Received and Metastatic Renal Cell Carcinoma (mRCC) Diagnosis
Description: In this outcome measure the duration form last treatment received including: partial nephrectomy, radical nephrectomy, radiation therapy, neoadjuvant systemic therapy and adjuvant systemic therapy was reported.
Time Frame: From last treatment received to mRCC diagnosis, during data identification period of 5 years (data recorded during approximately 12 months of retrospective observation period)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Months
Arm/Group | Sunitinib: Switched From 4/2 to 2/1 Schedule | Sunitinib 2/1 Schedule
Number analyzed (Participants) | 25 | 7
Months | 46.0 (50.3) | 59.1 (94.3)

14. Primary Outcome: Number of Systemic Lines of Treatment Received After the Diagnosis of Metastatic Renal Cell Carcinoma (mRCC)
Description: Number of participants were classified and reported according to the number of treatment lines received including first-line, second-line and third-line or more after diagnosis of mRCC.
Time Frame: From date of metastatic diagnosis to end of data identification period, for a maximum of 5 years (data recorded during approximately 12 months of retrospective observation period)
Population: Analysis population included all eligible participants whose data were retrieved from medical records and assessed.
Measure: Count of Participants; unit: Participants
Arm/Group | Sunitinib: Switched From 4/2 to 2/1 Schedule | Sunitinib 2/1 Schedule
Number analyzed (Participants) | 42 | 15
Participants
  First -line treatment | 15 | 14
  Second-line treatment | 20 | 0
  Three or more lines of treatment | 7 | 1

15. Primary Outcome: Duration of Each Systemic Lines of Treatment Received After the Diagnosis of Metastatic Renal Cell Carcinoma (mRCC)
Description: This outcome measure was analyzed by using Kaplan-Meier method.
Time Frame: Duration between initiating and termination date of each treatment line received after mRCC diagnosis, during data identification period of 5 years (data recorded during approximately 12 months of retrospective observation period)
Population: as for outcome 9
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Sunitinib: Switched From 4/2 to 2/1 Schedule | Sunitinib 2/1 Schedule
Number analyzed (Participants) | 42 | 15
Months
  First-line treatment | 12.3 [10.0 to 14.0] | 37.5 [7.5 to NA] — Upper limit for 95% CI could not be estimated because there were insufficient number of participants with event.
  Second-line treatment: number analyzed (Participants) | 27 | 1
  Second-line treatment | 6.5 [5.0 to 9.9] | NA [NA to NA] — Median and 95% CI could not be estimated because there were insufficient number of participants with event.
  Third-line treatment: number analyzed (Participants) | 7 | 1
  Third-line treatment | 6.6 [2.9 to NA] — Upper limit for 95% CI could not be estimated because there were insufficient number of participants with event. | NA [NA to NA] — Median and 95% CI could not be estimated because there were insufficient number of participants with event.

16. Primary Outcome: Duration of Treatment With Sunitinib
Time Frame: Day 1 of sunitinib first line treatment to end date of sunitinib treatment, during data identification period of 5 years (data recorded during approximately 12 months of retrospective observation period)
Population: Analysis population included all eligible participants whose data were retrieved from medical records and assessed. Data for this outcome measure is reported for evaluable participants in all of three arms including 4/2 schedule, 4/2 to 2/1 schedule and 2/1 schedule.
Measure: Mean (Standard Deviation); unit: Months
Groups:
- Sunitinib: Switched From 4/2 to 2/1 Schedule (4/2 Schedule): Participants with mRCC who initiated first-line treatment with sunitinib 50 mg per day on 4/2 schedule in the daily clinical practice, between 1-Jan-2014 and 30-Jun-2018 (+/- 6 months) were observed retrospectively over a duration of approximately 12 months.
Arm/Group | Sunitinib: Switched From 4/2 to 2/1 Schedule (4/2 Schedule) | Sunitinib: Switched From 4/2 to 2/1 Schedule | Sunitinib 2/1 Schedule
Number analyzed (Participants) | 42 | 42 | 15
Months | 4.6 (3.7) | 7.5 (5.5) | 13.6 (11.2)

17. Primary Outcome: Duration Between Discontinuation of 4/2 Schedule and Initiation of 2/1 Schedule
Time Frame: End date of 4/2 sunitinib schedule and start date of 2/1 sunitinib schedule, during data identification period of 5 years (data recorded during approximately 12 months of retrospective observation period)
Population: Analysis population included all eligible participants whose data were retrieved from medical records and assessed. Here, 'overall number of participants analyzed' signifies number of participants evaluable for this outcome measure.Data for this outcome measure is reported for evaluable participants in arm 4/2 to 2/1 schedule only.
Measure: Mean (Standard Deviation); unit: Months
Arm/Group | Sunitinib: Switched From 4/2 to 2/1 Schedule
Number analyzed (Participants) | 42
Months | 0.6 (0.7)

18. Primary Outcome: Participants With Reasons for Switching to 2/1 Treatment Schedule
Description: Number of participants with their reasons for switching to 2/1 schedule treatment including adverse event, local or professional protocol, participant decision, performance status and other (renal function deterioration; medical decision, site of cytoreductive surgery), were reported. One participant could have multiple reasons to switch to 2/1 treatment schedule.
Time Frame: Index date, during data identification period of 5 years (data recorded during approximately 12 months of retrospective observation period)
Population: Analysis population included all eligible participants whose data were retrieved from medical records and assessed. Data for this outcome measure is reported for evaluable participants in arm including 4/2 schedule only.
Measure: Count of Participants; unit: Participants
Arm/Group | Sunitinib: Switched From 4/2 to 2/1 Schedule (4/2 Schedule)
Number analyzed (Participants) | 42
Participants
  Adverse event | 31
  Local or professional protocol | 2
  Participant decision | 1
  Performance status | 10
  Other: Renal function deterioration | 1
  Other: Medical decision, site of cytoreductive surgery | 1
  Unknown | 3

19. Primary Outcome: Duration of Sunitinib 2/1 Treatment Schedule After Switching From 4/2 Treatment Schedule
Time Frame: From index date to end date of 2/1 treatment schedule, during data identification period of 5 years (data recorded during approximately 12 months of retrospective observation period)
Population: Analysis population included all eligible participants whose data were retrieved from medical records and assessed. Here, 'overall number of participants analyzed' signifies number of participants evaluable for this outcome measure. Data for this outcome measure is reported for evaluable participants in arms including 4/2 to 2/1 schedule only.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Sunitinib: Switched From 4/2 to 2/1 Schedule
Number analyzed (Participants) | 42
Months | 6.7 [6.0 to 10.3]

20. Primary Outcome: Number of Participants With Reasons for Sunitinib 2/1 Treatment Schedule Discontinuation
Description: Participants who had a termination of sunitinib treatment for reasons other than regimen change or switch, disease progression, or death were reported as discontinued. Categories with at least 1 non-zero data are reported below. One participant could have more than 1 reason for discontinuation.
Time Frame: From index date to end date of sunitinib 2/1 schedule, during data identification period of 5 years (data recorded during approximately 12 months of retrospective observation period)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Sunitinib: Switched From 4/2 to 2/1 Schedule | Sunitinib 2/1 Schedule
Number analyzed (Participants) | 38 | 9
Participants
  Adverse event | 4 | 0
  Participant decision | 2 | 1
  Progressive disease | 26 | 2
  Performance status | 1 | 0
  Lost to follow-up | 2 | 0
  Death | 3 | 2
  Unknown | 1 | 1
  Other | 2 | 3

21. Primary Outcome: Number of Participants With At-least 1 Dose Change
Time Frame: as for outcome 18
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | Sunitinib: Switched From 4/2 to 2/1 Schedule (4/2 Schedule) | Sunitinib: Switched From 4/2 to 2/1 Schedule | Sunitinib 2/1 Schedule
Number analyzed (Participants) | 42 | 42 | 15
Participants | 4 | 3 | 2

22. Primary Outcome: Number of Participants With Reason For Dose Change
Description: Participants who had change in the dose of sunitinib during the data identification period were reported. Categories with at least 1 non-zero data are reported below.
Time Frame: as for outcome 18
Population: Analysis population included all eligible participants whose data were retrieved from medical records and assessed. Here, 'overall number of participants analyzed' signifies number of participants evaluable for this outcome measure. Data for this outcome measure is reported for evaluable participants in all of three arms including 4/2 schedule, 4/2 to 2/1 schedule and 2/1 schedule.
Measure: Count of Participants; unit: Participants
Arm/Group | Sunitinib: Switched From 4/2 to 2/1 Schedule (4/2 Schedule) | Sunitinib: Switched From 4/2 to 2/1 Schedule | Sunitinib 2/1 Schedule
Number analyzed (Participants) | 4 | 3 | 2
Participants
  Adverse event | 4 | 3 | 2
  Adherence | 2 | 0 | 0

23. Primary Outcome: Number of Participants With Investigator Assessed Best Response to Treatment With Sunitinib
Description: Best response includes complete response (CR): equal to disappearance of all target lesions; partial response (PR): greater than equal to (>=) 30% decrease in sum of longest dimensions of lesions taking as reference baseline sum longest dimensions; progressive disease (PD): >=20% increase in sum of longest dimensions of lesions taking as a reference smallest sum of the longest dimensions since treatment start, or the appearance of >=1 new lesion; stable disease (SD): neither shrinkage for PR or increase for PD taking as reference smallest sum of longest dimensions since treatment start; as well as response not assessed and unknown also reported.
Time Frame: Index date up to end of follow up, disease progression, death, whichever occurred first during data identification period of 5 years (data recorded during approximately 12 months of retrospective observation period)
Population: Analysis population included all eligible participants whose data were retrieved from medical records and assessed.
Measure: Count of Participants; unit: Participants
Arm/Group | Sunitinib: Switched From 4/2 to 2/1 Schedule | Sunitinib 2/1 Schedule
Number analyzed (Participants) | 42 | 15
Participants
  Complete response | 4 | 4
  Partial response | 14 | 5
  Stable disease | 17 | 2
  Progressive disease | 5 | 3
  Response not assessed | 2 | 0
  Unknown | 0 | 1

24. Primary Outcome: Number of Participants With Different Supportive Care Elements During First Line Sunitinib Treatment
Description: Number of participants with different supportive care including anticoagulants, antibiotics, antidepressants, antidiarrheal, antiemetics, antifungals, antihistamines, antihypertensive medication, erythropoiesis stimulating agents (ESAs), granulocyte colony-stimulating factor (GSCF), hormone replacement, iron supplements, nutritional supplements, pain medications, platelet transfusion, red blood cell transfusion, steroids, topical skin care lotions/creams/moisturizers, other (pantoprazole) were reported. One participant could have more than 1 supportive care elements.
Time Frame: as for outcome 18
Population: Analysis population included all eligible participants whose data were retrieved from medical records and assessed. Data for this outcome measure is reported for evaluable participants in arms including 4/2 schedule only.
Measure: Count of Participants; unit: Participants
Arm/Group | Sunitinib: Switched From 4/2 to 2/1 Schedule (4/2 Schedule)
Number analyzed (Participants) | 42
Participants
  Anticoagulants | 3
  Antibiotics | 4
  Antidepressants | 4
  Antidiarrheal | 26
  Antiemetics | 14
  Antifungals | 2
  Antihistamines | 1
  Antihypertensive medication | 24
  ESAs | 2
  GSCF | 1
  Hormone replacement | 5
  Iron supplements | 4
  Nutritional supplements | 4
  Pain medications | 21
  Platelet transfusion | 0
  Red blood cell transfusion | 2
  Steroids | 3
  Topical skin care lotions/creams/moisturizers | 14
  Other: Pantoprazole | 1

25. Primary Outcome: Adverse Events Observed During First-line Treatment With Sunitinib
Description: An adverse event (AE) was any untoward medical occurrence in a participant who received investigational product without regard to possibility of causal relationship. AE was assessed according to severity; mild (not causing any significant problem, dose adjustment not required), moderate (caused problem that does not interfere significantly with usual activities or the clinical status, dose adjustment needed due to adverse event) and severe (caused problem that interferes significantly with usual activities or the clinical status, study drug stopped due to adverse event).
Time Frame: Day 1 of sunitinib first line treatment to follow up, during data identification period of 5 years (data recorded during approximately 12 months of retrospective observation period)
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | Sunitinib: Switched From 4/2 to 2/1 Schedule (4/2 Schedule) | Sunitinib: Switched From 4/2 to 2/1 Schedule | Sunitinib 2/1 Schedule
Number analyzed (Participants) | 42 | 42 | 15
Participants
  Mild | 42 | 42 | 14
  Moderate | 30 | 24 | 11
  Severe | 7 | 5 | 0

26. Primary Outcome: Progression Free Survival (PFS) From Initial Metastatic Diagnosis
Description: Progression free survival (PFS) was based on Kaplan-Meier estimates. PFS was defined as time in months from start of treatment-to-treatment discontinuation due to disease progression as assessed by the investigator. PD: =>20% increase in sum of longest dimensions of lesions taking as a reference smallest sum of longest dimensions since treatment start or appearance of =>1 new lesions. Disease progression was determined from oncologic assessment data (where data meet the criteria for PD), or from death case report forms (CRFs). This outcome measure was analyzed by using Kaplan-Meier method.
Time Frame: From date of mRCC diagnosis to date of disease progression, during data identification period of 5 years (data recorded during approximately 12 months of retrospective observation period)
Population: Analysis population included all eligible participants whose data were retrieved from medical records and assessed.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Sunitinib: Switched From 4/2 to 2/1 Schedule | Sunitinib 2/1 Schedule
Number analyzed (Participants) | 42 | 15
Months | 19.1 [15.0 to 25.2] | NA [17.2 to NA] — Median and upper limit of 95% CI were not estimable due insufficient number of participants with event.

27. Primary Outcome: Progression Free Survival (PFS) From Initiation of Sunitinib 4/2 Treatment Schedule
Description: PFS was based on Kaplan-Meier estimates. PFS was defined as time in months from start of treatment-to-treatment discontinuation due to disease progression as assessed by the investigator. PD: =>20% increase in sum of longest dimensions of lesions taking as a reference smallest sum of longest dimensions since treatment start or appearance of =>1 new lesions. Disease progression was determined from oncologic assessment data (where data meet the criteria for PD), or from death CRFs. This outcome measure was analyzed by using Kaplan-Meier method.
Time Frame: From date of initiation of sunitinib 4/2 schedule to date of disease progression, during data identification period of 5 years (data recorded during approximately 12 months of retrospective observation period)
Population: as for outcome 18
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Sunitinib: Switched From 4/2 to 2/1 Schedule (4/2 Schedule)
Number analyzed (Participants) | 42
Months | 16.6 [12.5 to 23.0]

28. Primary Outcome: Progression Free Survival (PFS) From Initiation of Sunitinib 2/1 Treatment Schedule
Description: as for outcome 27
Time Frame: From index date to date of disease progression, during data identification period of 5 years (data recorded during approximately 12 months of retrospective observation period)
Population: Analysis population included all eligible participants whose data were retrieved from medical records and assessed.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Sunitinib: Switched From 4/2 to 2/1 Schedule | Sunitinib 2/1 Schedule
Number analyzed (Participants) | 42 | 15
Months | 12 [6.5 to 17.7] | NA [16.0 to NA] — Median and Upper limit of 95% CI were not estimable due insufficient number of participants with event

29. Primary Outcome: Overall Survival (OS) From Metastatic Diagnosis
Description: Overall survival (OS) was defined as the time from the start of treatment to the date of death due to any cause. If a participant was not known to have died, survival was censored at the date of last known date participant alive. Kaplan-Meier method was used for OS analysis. This outcome measure was analyzed by using Kaplan-Meier method.
Time Frame: as for outcome 26
Population: Analysis population included all eligible participants whose data were retrieved from medical records and assessed.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Sunitinib: Switched From 4/2 to 2/1 Schedule | Sunitinib 2/1 Schedule
Number analyzed (Participants) | 42 | 15
Months | 46.1 [31.5 to NA] — Upper limit of 95% CI was not estimable due insufficient number of participants with event. | NA [22.6 to NA] — Median and upper limit of 95% CI were not estimable due insufficient number of participants with event.

30. Primary Outcome: Overall Survival (OS) From Initiation of Sunitinib 4/2 Treatment Schedule
Description: OS was defined as the time from the start of treatment to the date of death due to any cause. If a participant was not known to have died, survival was censored at the date of last known date participant alive. Kaplan-Meier method was used for OS analysis. This outcome measure was analyzed by using Kaplan-Meier method.
Time Frame: as for outcome 26
Population: Analysis population included all eligible participants whose data were retrieved from medical records and assessed. Data for this outcome measure is reported for evaluable participants in arm including 4/2 to 2/1 schedule only.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Sunitinib: Switched From 4/2 to 2/1 Schedule
Number analyzed (Participants) | 42
Months | 46.1 [29.1 to NA] — Upper limit of 95% CI was not estimable due insufficient number of participants with event.

31. Primary Outcome: Overall Survival (OS) From Initiation of Sunitinib 2/1 Treatment Schedule
Description: as for outcome 30
Time Frame: as for outcome 26
Population: Analysis population included all eligible participants whose data were retrieved from medical records and assessed.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Sunitinib: Switched From 4/2 to 2/1 Schedule | Sunitinib 2/1 Schedule
Number analyzed (Participants) | 42 | 15
Months | 42.0 [26.0 to NA] — Upper limit of 95% CI was not estimable due insufficient number of participants with event. | NA [16.5 to NA] — Median and upper limit of 95% CI were not estimable due insufficient number of participants with event.

32. Primary Outcome: Time to Initiate Second Line Treatment
Time Frame: From mRCC diagnosis to start date of second line treatment and from end date of first line treatment to start date of second line treatment,data identification period of 5 years(data recorded during approx. 12 months of retrospective observation period)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Months
Arm/Group | Sunitinib: Switched From 4/2 to 2/1 Schedule | Sunitinib 2/1 Schedule
Number analyzed (Participants) | 27 | 1
Months
  From mRCC diagnosis | 19.7 (16.4) | 37.5 (NA) — Standard deviation was not estimable due insufficient number of participants with event.
  From first-line discontinuation | 2.6 (2.9) | 28.0 (NA) — Standard deviation was not estimable due insufficient number of participants with event.

ADVERSE EVENTS:
Time Frame: From 01-Jan-2014 to 30-Jun-2018 (+/- 6 months), for a maximum of 5 years (data recorded during 12 months of retrospective observation period)
Description: Same event may appear as both an AE and a serious AE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another participant, or one participant may have experienced both a serious and non-serious event during the study. No source vocabulary name used for adverse event reporting', because of the retrospective nature of the study and physicians were asked to report evidence of AE as: mild, moderate, or severe.
Arm/Group | Sunitinib: Switched From 4/2 to 2/1 Schedule (4/2 Schedule) | Sunitinib: Switched From 4/2 to 2/1 Schedule | Sunitinib 2/1 Schedule
All-Cause Mortality (participants affected / at risk) | 0/42 | 20/42 | 3/15
Serious Adverse Events (participants affected / at risk) | 7/42 | 5/42 | 0/15
Other Adverse Events (participants affected / at risk) | 42/42 | 42/42 | 14/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sunitinib: Switched From 4/2 to 2/1 Schedule (4/2 Schedule) (N=42) | Sunitinib: Switched From 4/2 to 2/1 Schedule (N=42) | Sunitinib 2/1 Schedule (N=15)
Mucositis (Gastrointestinal disorders) | 2 | 0 | 0
Asthenia (General disorders) | 3 | 2 | 0
Fatigue (General disorders) | 4 | 3 | 0
Pain (General disorders) | 0 | 1 | 0
Stomatitis (General disorders) | 0 | 1 | 0
Dysgeusia (Nervous system disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 3 | 2 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Hand and foot syndrome (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Anemia (Blood and lymphatic system disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sunitinib: Switched From 4/2 to 2/1 Schedule (4/2 Schedule) (N=42) | Sunitinib: Switched From 4/2 to 2/1 Schedule (N=42) | Sunitinib 2/1 Schedule (N=15)
Diarrhea (Gastrointestinal disorders) | 31 | 33 | 10
Dry mouth (Gastrointestinal disorders) | 12 | 13 | 10
Dyspepsia (Gastrointestinal disorders) | 17 | 13 | 3
Mucositis (Gastrointestinal disorders) | 22 | 25 | 4
Nausea (Gastrointestinal disorders) | 18 | 15 | 11
Vomiting (Gastrointestinal disorders) | 8 | 9 | 4
Asthenia (General disorders) | 35 | 31 | 9
Changes in hair color (General disorders) | 15 | 11 | 6
Chills (General disorders) | 1 | 3 | 1
Fatigue (General disorders) | 16 | 17 | 9
Influenza-like illness (General disorders) | 1 | 2 | 1
Pain (General disorders) | 18 | 14 | 4
Pyrexia (General disorders) | 2 | 4 | 0
Stomatitis (General disorders) | 14 | 12 | 3
Anorexia (Metabolism and nutrition disorders) | 21 | 18 | 8
Dysgeusia (Nervous system disorders) | 13 | 13 | 0
Headache (Nervous system disorders) | 3 | 6 | 5
Hypertension (Vascular disorders) | 23 | 23 | 6
Hypothyroidism (Endocrine disorders) | 10 | 12 | 3
Heart failure (Cardiac disorders) | 0 | 3 | 1
Decline in ejection fraction (Cardiac disorders) | 2 | 4 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 11 | 16 | 6
Hand and foot syndrome (Skin and subcutaneous tissue disorders) | 21 | 19 | 7
Rash (Skin and subcutaneous tissue disorders) | 2 | 4 | 4
Skin discoloration (Skin and subcutaneous tissue disorders) | 11 | 9 | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 10 | 7 | 8
Neutropenia (Blood and lymphatic system disorders) | 5 | 7 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 7 | 4 | 4
Leukopenia (Blood and lymphatic system disorders) | 8 | 6 | 1
Anemia (Blood and lymphatic system disorders) | 18 | 18 | 5
Lymphopenia (Blood and lymphatic system disorders) | 5 | 3 | 1
Liver toxicity (Hepatobiliary disorders) | 2 | 1 | 1
Renal toxicity (Renal and urinary disorders) | 1 | 5 | 2
CPK increased (Investigations) | 4 | 1 | 2
Lipase increased (Investigations) | 6 | 2 | 2
Aspartate aminotransferase increased (Investigations) | 6 | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-13): https://cdn.clinicaltrials.gov/large-docs/89/NCT04115189/Prot_SAP_000.pdf